CLINICAL TRIAL: NCT03363347
Title: Association Between BRAF V600E and Redifferentiation Therapy in Patients With Radioiodine-refractory Papillary Thyroid Cancer
Brief Title: BRAF V600E and Redifferentiation Therapy in Radioiodine-refractory Papillary Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Stefan Kopf MD, Head of the Clinical Study Center for Diabetes Research, Heidelberg University
Other Study IDs: S-206/2005
Record Dates: First submitted 2017-11-20; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radioiodine refractory papillary thyroid cancer: Patients with radioiodine refractory papillary thyroid cancer who received redifferentiation therapy with retinoid acid.
  Interventions: Drug: Redifferentiation with retinoid acid
- Radioiodine sensitive papillary thyroid cancer: Patients who were in remission after one or two radioiodine therapies.

INTERVENTIONS:
Drug: Redifferentiation with retinoid acid — In this retrospective study, patients with radioiodine refractory papillary thyroid cancer routinely received (clinical indication, no study medication was given) retinoid acid for redifferentiation prior to further course of radioiodine therapy.
  Groups: Radioiodine refractory papillary thyroid cancer

SUMMARY:
Papillary thyroid cancer (PTC) is the most common neoplasia in the thyroid gland. The combination of surgery, followed by radioiodine therapy (RIT) and thyroid-stimulating hormone (TSH) suppressive therapy is usually a curative option for differentiated thyroid cancer (DTC). Although DTC has a good prognosis generally, it is problematic when dedifferentiation is suspected and radioiodine refractoriness presumed. One possible therapy option for redifferentiation is the pretreatment with retinoids. From 2008 to 2014 there were 13 patients with PTC who were treated with retinoids after thyroidectomy before a further course of radioiodine. A recent study has shown that the efficacy of Selumetinib, another option for redifferentiation depends on the mutational status of the treated patient. In this retrospective study the investigators looked for a similar association between BRAF V600E and redifferentiation therapy with retinoids. As retinoids have fewer side effects compared to TKI, it is worth performing studies to assess the importance of genetic marker for the response and to estimate the chances of this specific patient collective. BRAF V600E seems to be associated with better long-term response after redifferentiation therapy with 13-cis RA in RAI-R PTC. Therefore, evaluation of BRAF mutational status prior to redifferentiation therapy could be beneficial for predicting response.

ELIGIBILITY:
Eligible criteria for radioiodine-refractory patients included:

* PTC
* no response to former RIT
* decrease or loss of initial sufficient RI-Uptake
* redifferentiation therapy with 13-cis-RA
* available FFPE tissue.

Eligible criteria for radioiodine-sensitive patients included:

* PTC
* cured after a maximum of two RIT
* no redifferentiation therapy necessary
* available FFPE tissue.

Exclusion criteria

* DTC other than PTC
* patients lost to follow-up
* other redifferentiation therapy than retinoids
* anaplastic or medullary thyroid cancer
* benign thyroid disease, no available FFPE tissue
* more than two RITs in the control group
* insufficient clinical information.

Ages: 24 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twelve patients with radioiodine-refractory papillary thyroid cancer were treated with retinoic acid before a further course of radioiodine therapy. One patient had to be excluded from the analysis due to missing data in this retrospective analysis. Furthermore, they were compared with twelve patients with radioiodine-sensitive thyroid cancer who were considered as cured after a maximum of two radioiodine therapies.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Response to radioiodine therapy after redifferentiation | 7 years
  Redifferentiation therapy was performed using 13-cis RA (Isotretinoin, Roaccutan®) with a daily dose of orally 1,5mg/kg for up to two months. For assessment of clinical outcome of 13-cis retinoic acid treatment three parameters, tumor size, thyroglobulin levels and radioiodine uptake were considered in a graduated model.

SECONDARY OUTCOMES:
Parameter tumor size | 7 years
  Tumor size was evaluated form CT, MRI, or FDG-PET/CT imaging, comparing results before and after redifferentiation and RIT, results were evaluated using Response Evaluation Criteria in Solid Tumors (RECIST).
Parameter thyroglobulin levels (serum Tg) | 7 years
  Non-stimulated serum Tg level (in ng/ml) before redifferentiation therapy was compared with the first Tg level after redifferentiation and RIT. A stable Tg level was defined as ≤10% difference.
Parameter radioiodine-uptake (RI-Uptake) | 7 years
  Recovery of RI-Uptake was evaluated from the post-therapy whole body scan in comparison to the lesions in CT, MRI, or FDG-PET/CT imaging before redifferentiation. Optimal uptake was defined as intensive accumulation of radioiodine in all tumor lesions. When not all lesions accumulate radioiodine or the signal was weak it was considered as suboptimal uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kopf, MD, Principal Investigator — Head of the Clinical Study Center for Diabetes Research

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03363347/Prot_000.pdf